CLINICAL TRIAL: NCT06356519
Title: Effectiveness and Safety of Sacituzumab Govitecan in Chinese Metastatic Breast Cancer: A Multi-center Real-world Retrospective Study
Brief Title: Real-world Effectiveness and Safety Study of Sacituzumab Govitecan in Chinese Metastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-29
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Sacituzumab Govitecan; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacituzumab Govitecan: Sacituzumab Govitecan,10 mg/kg ivgtt d1, d8, q3w
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan,10 mg/kg ivgtt d1, d8, q3w

SUMMARY:
The aim of this trial is to explore the real-world effectiveness and poteintial predictors of Sacituzumab Govitecan in Chinese metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old.
2. Metastatic breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
3. Plan to receive or has received Sacituzumab Govitecan monotherapy
4. Available medical history.

Exclusion Criteria:

1. Incomplete medical history.
2. Pregnancy or breast-breeding

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years old with metastatic breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
ORR | 6 weeks
  Overall Response Rate
OS | 6 weeks
  Overall Survival
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 6 weeks
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China